CLINICAL TRIAL: NCT05562271
Title: A Multi-center, Randomized, Single-blinded, Exploratory Clinical Trial to Evaluate Safety and Efficacy of Alleviating Symptom of Low-dose RaDiation Therapy in Patients With KNee osteoArthritis
Brief Title: Clinical Trial of Low-dose Radiation Therapy in Patients With Knee Osteoarthritis (LoRD-KNeA Trial)
Acronym: LoRD-KNeA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); SMG-SNU Boramae Medical Center (Other); Korea Hydro & Nuclear Power (Unknown)
Responsible Party: Principal Investigator, Byoung Hyuck Kim, Prof. Dr., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N22S005000
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee; Osteoarthritis; radiation therapy; radiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- sham radiation therapy (Sham Comparator): sham radiation therapy
  Interventions: Radiation: sham radiation therapy
- low-dose radiation therapy, 30 cGy/6 fx (experimental 1) (Experimental): low-dose radiation therapy, 30 cGy/6 fx
  Interventions: Radiation: low-dose radiation therapy
- low-dose radiation therapy, 300 cGy/6 fx (experimental 2) (Experimental): low-dose radiation therapy, 300 cGy/6 fx
  Interventions: Radiation: low-dose radiation therapy

INTERVENTIONS:
Radiation: low-dose radiation therapy — low-dose radiation therapy to involved knee joint
  Arms: low-dose radiation therapy, 30 cGy/6 fx (experimental 1); low-dose radiation therapy, 300 cGy/6 fx (experimental 2)
Radiation: sham radiation therapy — sham radiation therapy to involved knee joint
  Arms: sham radiation therapy

SUMMARY:
Clinical verification of knee osteoarthritis pain relief and functional improvement using low-dose radiation therapy

DETAILED DESCRIPTION:
This clinical trial is a multicenter, randomized, single-blinded, exploratory clinical trial to evaluate the efficacy and safety of low-dose radiation for knee osteoarthritis patients. The experimental group is treated with low-dose irradiation 6 times for 3 weeks according to the dose determined for each group, and the control group is treated with sham irradiation. Both the experimental group and the control group visit the hospital 4 weeks after irradiation and at 4, 8, and 12 months to evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-85 years old
* Kellgren-Lawrence grade 2-3 and diagnosed as a patient with primary knee osteoarthritis according to the ACR knee OA diagnostic criteria
* Patients with VAS 40 or higher when walking, with or without medication at the time of screening
* Patients who have VAS 50 or more and 90 or less when walking at the baseline
* Among patients who were previously taking analgesic drugs at the time of screening, those with an increase in pain of 10 points or more at the baseline
* Patients who do not want to take non-narcotic analgesics, those who have failed to control their pain due to the use of non-narcotic analgesics, or candidates for invasive treatment (intra-articular injection, arthroplasty, etc.)
* A person who has a will to discontinue all pain medications except for rescue medications throughout screening, baseline, and clinical trials related to knee arthritis
* A person who gives consent to use an approved contraceptive method from screening to 3 months after the end of the clinical trial
* A person who understands the eligibility requirements for the study and has signed the consent form

Exclusion Criteria:

* A history of knee irradiation in the past
* Patients participating in other degenerative arthritis clinical trials
* Kellgren-Lawrence grade 4
* A history of malignancy within the last 5 years
* A history of knee or hip surgery in the past
* Patients who have received systemic steroid treatment or intra-articular steroid/hyaluronic acid injection within 2 months of screening
* Patients with hip degenerative arthritis or other diseases of NRS 5 or higher that may affect functional score evaluation
* Patients who are scheduled for surgical treatment of the knee joint during the clinical trial period
* BMI > 39 kg/m2
* Known history of analgesic or substance abuse within 2 years of screening
* History, diagnostic signs or symptoms of any of the following clinically significant psychiatric disorders that would render the study ineligible (psychotic disorder, depression, somatic disorder)
* History, diagnostic signs, or symptoms of any of the following clinically significant heart diseases that would render the study ineligible (surgery or stenting for ischemic heart disease and coronary artery disease within 6 months prior to screening)
* History of other diseases that may affect the index joint, including autoimmune diseases (lupus, rheumatoid arthritis, etc.)
* Fibromyalgia history or diagnosis
* If the researcher judges that a person with significant trauma or other findings considered clinically important is inappropriate for participation in this study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
OMERACT-OARSI response rate | 4 months
  OMERACT-OARSI (Outcome Measures in Rheumatology-Osteoarthritis Research Society International) response rate at 4 months. The OMERACT-OARSI criteria for response are (1) improvement in pain or physical function ≥50% and an absolute change ≥20 mm; or (2) improvement of ≥20% with an absolute change ≥10 mm in at least two of the following three categories: pain, physical function, and patient's global assessment.

SECONDARY OUTCOMES:
OMERACT-OARSI response rate | 4 weeks, 8 months, 12 months
  OMERACT-OARSI (Outcome Measures in Rheumatology-Osteoarthritis Research Society International) response rate at 4 weeks, 8 months, and 12 months. The OMERACT-OARSI criteria for response are (1) improvement in pain or physical function ≥50% and an absolute change ≥20 mm; or (2) improvement of ≥20% with an absolute change ≥10 mm in at least two of the following three categories: pain, physical function, and patient's global assessment.
Changes in WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) score | 4 weeks, 4 months, 8 months, 12 months
  Total score (min 0, max 96 points, higher scores mean a worse outcome) and WOMAC score subscale (pain: min 0 max 20, stiffness: min 0 max 8, physical function: min 0 max 68)
Changes in pain score | 4 weeks, 4 months, 8 months, 12 months
  VAS score (min 0, max 100, higher scores mean a worse outcome)
Changes in global assessment | 4 weeks, 4 months, 8 months, 12 months
  PGA (Patient Global Assessment) score (min 0, max 100, higher scores mean a worse outcome)
Radiological Changes Evaluated by Knee MRI | 4 months, 12 months
  Radiological Changes Evaluated by Knee MRI
Radiological Changes Evaluated by Knee X-ray | 12 months
  Radiological Changes Evaluated by Knee X-ray
Changes in serum ESR (Erythrocyte sedimentation rate) | 4 weeks, 4 months, 8 months, 12 months
  Changes in ESR (Erythrocyte sedimentation rate)
Changes in serum CRP (C-reactive protein) | 4 weeks, 4 months, 8 months, 12 months
  Changes in CRP (C-reactive protein)
Change in the amount of analgesic rescue medication usage | 4 weeks, 4 months
  Concomitant use of analgesics is prohibited until 4 months after irradiation, when the primary efficacy evaluation is scheduled. During this period, the use of a rescue drug (acetaminophen) may be permitted if the subjects need it for osteoarthritis. Monitor the amount of rescue medication prescribed to measure changes in usage during visits up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Hyuck Kim, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (3):
- South Korea (3):
  - Seoul National University Hospital / SMG-SNU Boramae Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim BH, Shin K, Kim MJ, Kim HJ, Ro DH, Wang JH, Lee DH, Kim DH, Sun J, Lee JH, Kim JY, Hong EH, Cho SJ, Han HS, Park W. Low-dose RaDiation therapy for patients with KNee osteoArthritis (LoRD-KNeA): a protocol for a sham-controlled randomised trial. BMJ Open. 2023 Feb 10;13(2):e069691. doi: 10.1136/bmjopen-2022-069691. PMID 36764712